CLINICAL TRIAL: NCT03468036
Title: Intratracheal Suctioning and Oxygenation at Extubation (INnovATE)
Brief Title: Intratracheal Suctioning and Oxygenation at Extubation
Acronym: INNOVATE
Status: Completed | Type: Observational
Sponsor: Jörg Schefold (Other)
Responsible Party: Sponsor-Investigator, Jörg Schefold, Sponsor-investigator, Insel Gruppe AG, University Hospital Bern
Organization: Insel Gruppe AG, University Hospital Bern (Other)
Other Study IDs: INNOVATE
Record Dates: First submitted 2018-03-09; First posted 2018-03-16 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Extubation
Keywords: critical illness; ICU; extubation; respiratory failure
MeSH Terms: conditions — Critical Illness; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Extubation with 100% O2: for further information please refer to study protocol
  Interventions: Other: none, does not apply
- Extubation with 35% O2: for further information please refer to study protocol
  Interventions: Other: none, does not apply

INTERVENTIONS:
Other: none, does not apply — none: does not apply

SUMMARY:
Data analysis of routinely applied extubation procedures on the ICU: i.e. extubation with 100% O2 vs. 35% O2 with/without suctioning.

ELIGIBILITY:
Inclusion Criteria:

* All adult (≥18 years) ICU patients with routine extubation on the ICU during the 2-month observational interval.

Exclusion Criteria:

* Age < 18 years
* Patients on comfort therapy and/ or terminal extubation or accidental extubationtracheostomized patients
* Patients with refusal to general consent or withdrawal of general consent (DLF and/or internal database)
* Patients dying without next-of-kin available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients that undergo routine extubation
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Difference in proportion of patients with need for ongoing ventilatory support | 30 days max follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Joerg C Schefold, MD, Principal Investigator — Inselspital, University of Bern
Locations (1):
- Dept. of Intensive Care Medicine, University of Bern,, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided